CLINICAL TRIAL: NCT06537726
Title: Real-time Breath Analysis for the Detection of Invasive Fungal Infections in Neutropenic High-risk Patients
Brief Title: Breath Analysis for the Detection of Invasive Fungal Infections
Acronym: REDEFINE
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Jeremy Deuel, Principal Investigaor, University of Zurich
Other Study IDs: SNCTP000005947
Record Dates: First submitted 2024-07-27; First posted 2024-08-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Lymphoblastic; Neutropenia; Chemotherapy-induced Neutropenia; Invasive Fungal Infections; Invasive Pulmonary Aspergillosis
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neutropenia; Invasive Fungal Infections; Invasive Pulmonary Aspergillosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- No invasive fungal disease: Patients, that retrospectively do not have evidence of IFI
  Interventions: Diagnostic Test: Secondary electrospray ionization high-resolution mass spectrometry (SESI-HRMS)
- Possible invasive fungal disease: Patients, that retrospectively have a possible IFI (according to EORTC guidelines). There is suspicion of IFI by clinical or radiological features, but no microbiological evidence of IFI.
  Interventions: Diagnostic Test: Secondary electrospray ionization high-resolution mass spectrometry (SESI-HRMS)
- Probable invasive fungal disease: Patients, that retrospectively have a probable IFI (according to EORTC guidelines). There is suspicion of IFI by clinical or radiological features, and indirect microbiological evidence of IFI.
  Interventions: Diagnostic Test: Secondary electrospray ionization high-resolution mass spectrometry (SESI-HRMS)
- Proven invasive fungal disease: Patients, that retrospectively have a proven IFI (according to EORTC guidelines). There is histological (angioinvasive growth of a fungus) or definitive microbiological evidence of IFI, e.g. evidence of a fungus from a sterile tissue.
  Interventions: Diagnostic Test: Secondary electrospray ionization high-resolution mass spectrometry (SESI-HRMS)

INTERVENTIONS:
Diagnostic Test: Secondary electrospray ionization high-resolution mass spectrometry (SESI-HRMS) — Identify volatile biomarkers of IFI by analyzing the breath metabolome of patients with proven or probable IFI according to the criteria outlined by EORTC/MSG and controls.
  Other Names: Blood sampling (serologic biomarkers, PCR); Sputum analysis; Low-dose CT

SUMMARY:
Patients with leukemia and concomitant neutropenia are at high risk of developing invasive fungal infections (IFI) that are associated with high morbidity and mortality. As these patients typically have severe thrombocytopenia, direct diagnostic sampling with invasive procedures is often not possible due to the high peri-interventional risk. Therefore, the presumptive diagnosis of IFI is primarily based on compatible lung findings on computed tomography and serologic detection of fungal cell wall components, which, however, have limited sensitivity and specificity.

With the present study, the investigators aim to determine a set of specific volatile biomarkers in leukemia patients with proven or probable IFI using secondary electrospray ionization high-resolution mass spectrometry (SESI-HRMS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute leukemia
* Planned chemotherapy with a duration of hospitalisation of 2 weeks or longer
* Neutropenia (<500/µl) present at inclusion or planned chemotherapy with expected neutropenia (<500/µl) for more than 7 days

Exclusion Criteria:

* Unable to follow instructions for breath analysis
* Anatomic abnormalities precluding the use of a mouthpiece for breath analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute leukemia that are undergoing chemotherapy at the Department of Medical Oncology and Haematology at the University Hospital Zurich
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Novel biomarker (m/z value) for IFI by SESI-HRMS | through study completion, on average after 3 weeks
  Feature in Mass Spectrometry

SECONDARY OUTCOMES:
Specificity and sensitivity of this novel biomarker | through study completion, on average after 3 weeks
  Description of Accuracy and Precision of this novel biomarker
Anticipation of IFI | through study completion, on average after 3 weeks
  Timepoint of first detection in relation to first clinical symptoms of IFI

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Deuel, PD Dr., Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided